CLINICAL TRIAL: NCT03282773
Title: Optimal Strategy of Primary Percutaneous Coronary Intervention for Acute Myocardial Infarction Due to Unprotected Left Main Coronary Artery Occlusion
Brief Title: Optimal Strategy of Primary PCI for Left Main Coronary Artery Occlusion Induced AMI
Acronym: OPTIMAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-104
Record Dates: First submitted 2017-09-10; First posted 2017-09-14 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Acute Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: acute myocardial infarction; percutaneous coronary intervention; deferred stent implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferred stent implantation (Experimental): Drug-eluting stents are implanted 4-10 days after primary angiography and restoration of blood flow in left main coroanry artery in a secondary PCI
  Interventions: Device: Deferred stent implantation
- Immediate stent implantation (Active Comparator): Drug-eluting stents are implanted immediately after primary angiography and restoration of blood flow in left main coroanry artery
  Interventions: Device: Immediate stent implantation

INTERVENTIONS:
Device: Deferred stent implantation — Primary angiography and pretreatment including balloon dilatation and thrombus aspiration, second generation drug-eluting stents are implanted 4-10 days after restoration of blood flow in left main coronary artery in a secondary PCI.
  Arms: Deferred stent implantation
Device: Immediate stent implantation — Primary angiography and pretreatment including balloon dilatation and thrombus aspiration, second generation drug-eluting stents are implanted immediately after restoration of blood flow in left main coronary artery in a secondary PCI.
  Arms: Immediate stent implantation

SUMMARY:
This study will compare clinical outcomes of immediate stent implantation with deferred stent implantation(4-10days after primary angiography) for patients presented with acute myocardial infarction due to left main coronary artery occlusion.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention for patients presented with acute myocardial infarction caused by left main coronary artery occlusion is associated with significantly higher mortality and risks of major cardiac adverse events. Deferred stent implantation may improve prognosis of primary PCI through reducing distal embolization and no-reflow phenomenon. There is no randomized clinical trial focuses on the effect and outcome of deferred stent implantation on primary PCI for left main coronary artery occlusion in contrast with conventional strategy.

This prospective, multicenter, randomized trial is aimed to compare immediate stenting with deferred stenting for LM-AMI with 30 centers in China involved. We hope to determine whether deferred stenting is superior to conventional strategy for primary PCI of AMI caused by left main coronary artery occlusion in improving long-term clinical outcomes and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute myocardial infarction occured within 12 hours
* Left main coronary artery occlusion confirmed by angiography
* Left main coronary artery occlusion (TIMI flow 0,1 or 2) confirmed by primary angiography, TIMI flow grade 3 achieved after pretreatment of thrombus aspiration or balloon dilatation

Exclusion Criteria:

* Life expectancy less than 1 years
* Cardiogenic shock
* Chronic kidney disease, stage 4 by KDOQI(GFR<30ml/min)
* Contraindications to aspirin or other anti-platelet drugs
* Allergy to contrast agent, rapamycin or paclitaxel
* Patients who are included in other ongoing trials
* Pregnant female

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiac death and recurrent myocardial infarction | 30 days after primary angiography
  Recorded in follow-up

SECONDARY OUTCOMES:
All cause death, cardiac death, recurrent myocardial infarction, target vessel revascularization | 30 days after primary angiography
  Recorded in follow-up
Residual stenosis of left main coronary artery | Immediately after stent implantation and 12 months after primary angiography
  Measured through angiography
Left ventricular ejection fraction | 30 days and 12 months after primary angiography
  Measured through echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Principal Investigator — Zhongshan Hospital,Shanghai
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Gao Y, Zhang F, Li C, Dai Y, Yang J, Qu Y, Qian J, Ge J; OPTIMAL trial investigators. Optimal strategy of primary percutaneous coronary intervention for acute myocardial infarction due to unprotected left main coronary artery occlusion (OPTIMAL): study protocol for a randomised controlled trial. Trials. 2019 Mar 8;20(1):162. doi: 10.1186/s13063-019-3211-0. PMID 30850023